CLINICAL TRIAL: NCT04584775
Title: Implementing Acupuncture and Chinese Herbal Medicine Into Palliative Care: A Randomized Controlled Open-label Clinical Trial
Brief Title: Implementing Acupuncture and Chinese Herbal Medicine Into Palliative Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid19 Pandemia
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Palliach
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Advanced Cancer; Lung Cancer; Breast Cancer; Colo-rectal Cancer; Pancreas Cancer; Cholangiocarcinoma; Quality of Life; Symptoms and Signs
Keywords: Palliative Care; Traditional Chinese Medicine; Acupuncture; Chinese Herbal Medicine
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma; Signs and Symptoms | interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: Traditional Chinese Medicine plus Standard Care versus Standard Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine plus Standard Care (Experimental): Participants in this group will receive standard Palliative Care and will additionally see a practitioner of Traditional Chinese Medicine. No strict protocol for the actual intervention exists (pragmatic approach). The participants will at least receive acupuncture and/or chinese herbal medicine. The standard care will include any established medical intervention according to currently available guidelines in palliative care.
  Interventions: Other: Treatment modalities of Traditional Chinese Medicine (Acupuncture, Chinese herbal medicine, Tunia, Chinese dietetics); Other: Standard care
- Standard Care (Other): The standard care will include any established medical intervention according to currently available guidelines in palliative care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Treatment modalities of Traditional Chinese Medicine (Acupuncture, Chinese herbal medicine, Tunia, Chinese dietetics) — Acupuncture is a physical treatment modality that uses thin needles to stimulate specific points on the body in order to manipulate neurologic mechanisms to control specific symptoms and/or physiologic processes.
  Chinese herbal medicine is a phytotherapeutic treatment modality that uses herbs, minerals and rarely animal products which are orally administered.
  Tuina is a form of massage and physical therapy. Chinese dietetics is a nutritional therapy according to the theoretical principle of traditional Chinese medicine.
  Arms: Traditional Chinese Medicine plus Standard Care
Other: Standard care — Standard care includes any medical intervention in palliative care that aims to promote and/or sustain the quality of life of patients suffering from advanced disease (in this case cancer). These may be of pharmaceutical, surgical, psychological and/or spiritual nature.

SUMMARY:
In this clinical trial we want to investigate the clinical benefit of a complementary therapy using therapeutical modalities of the traditional chinese medicine in patients suffering from advanced cancer.

DETAILED DESCRIPTION:
After giving informed consent, the participants will be randomized into two groups (1:1). Both groups will receive standard care while one group will additionally be assigned to a practitioner of traditional Chinese medicine (TCM) who will deliver a individual treatment according to the needs of the participant (pragmatic approach).

Outcome measures will be monitored over the course of eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* One of the following tumor entities

  * Colorectal cancer (CRC)
  * Lung cancer (SCLC, NSCLC)
  * Breast cancer (BC)
  * Pancreas/Cholangiocellular cancer
* Best supportive care (i.e., no currently ongoing tumor-specific therapy)

  o Exception: palliative anti-hormonal therapy or palliative radiotherapy
* Performance status: ECOG 0 to 2
* Estimated life expectancy > 4 months

Exclusion Criteria:

* Any serious concomitant systemic disorder
* Pregnancy or breast-feeding
* Impossibility to attend TCM practices in Graz
* Incapacity to comply/consent
* Language barrier
* Brain metastases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in FACT-G at week 4 | Baseline and week 4
  FACT-G ((Functional Assessment of Cancer Therapy - General) is a validated multi-dimensional quality of life (QoL) questionnaire. It consists of 26 items and addresses four dimensions of QoL, including physical wellbeing (PWB), functional wellbeing (FWB), emotional wellbeing (EWB), and social wellbeing (SWB). The scoring system is a five-point Likert scale assessing the QoL of the past seven days. The FACT-G total score has a range of 0-108, whereas higher scores indicate a higher QoL.

SECONDARY OUTCOMES:
Change from baseline in FACT-G at week 8 | Baseline and week 8
  FACT-G is a validated multi-dimensional quality of life questionnaire. It consists of 26 items and addresses four dimensions of QoL, including physical wellbeing (PWB), functional wellbeing (FWB), emotional wellbeing (EWB), and social wellbeing (SWB). The scoring system is a five-point Likert scale assessing the QoL of the past seven days. The FACT-G total score has a range of 0-108, whereas higher scores indicate a higher QoL.
Change from baseline in PHQ-9 at week 4 and 8 | Baseline and week 4 and 8
  The PHQ-9 (Patient Health Questionnaire) aims at depressive disorders in medically ill populations. It is a 9-item diagnostic tool based upon the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders IV) criteria for major depressive disorder. The PHQ-9 score has a range of 0-27, whereas a score above 10 indicates major depression,
  This questionnaire will also be completed by a close caregiver (family or friend).
Change of symptom burden, assessed by ESAS-R | Baseline and weekly until week 8
  The ESAS-R (Edmonton Symptom Assessment Scale revised) was established specifically for palliative care patients and is a nine-item patient-rated symptom visual analog scale. Each item is rated by a numerical rating scale (0-10), whereas higher numbers indicate a more severe symptom experience. The total score of all symptoms represents the total symptom-burden, whereas a higher score indicates a higher total symptom-burden.
Change in use of Pro re nata medication (P.R.N.M.), assessed by Pro re nata medication diary | Daily from baseline to week 8
  To assess the use of pro re nata medication, the participants will document their usage in a diary. P.R.N.M. may be antiemetics, analgetics, tranquilizers or any other drug used for acute symptom relieve.
Change from baseline in FAMCARE-2 at week 4 and 8 | Baseline and week 4 and 8
  To evaluate the satisfaction of advanced cancer care in family or friends caregivers, the family satisfaction with end-of-life care two questionnaire (FAMCARE-2) will be used. It is a 17-item assessment tool using a Likert scale (score: 0-68), including subscales for information giving, physical patient care, psychosocial care, and availability of care. A high score on the FAMCARE-2 is associated with a high satisfaction with the palliative care service.
  This questionnaire will only be completed by a close caregiver (family or friend).

OTHER OUTCOMES:
Change from baseline in Performance Scales at week 4 and 8 | Baseline and week 4 and 8
  The Karnofsky Performance Scale describes a patient's ability to perform daily activities without restrictions due to disease through to death on a scale of 100 to 0, in steps of 10. Additionally, the ECOG (Eastern Cooperative Oncology Group) Performance Scale, which is a six-grade scale that assesses the level of functioning in terms of self-care, activity, and physical ability, will be assessed.
Number of consultations of the mobile palliative care team | From baseline to week 8
  Throughout the course of the study, the number of consultations of the mobile palliative care team will be documented and compared between the two groups.
Number of hospital referrals | From baseline to week 8
  Throughout the course of the study, hospital referrals will be documented and compared between the two groups.
Length of hospitalizations | From baseline to week 8
  Throughout the course of the study, the length of hospitalizations will be documented and compared between the two groups.
Overall survival | From baseline to week 8.
  All deaths throughout the course of the study will be documented to calculate the overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided